CLINICAL TRIAL: NCT01814189
Title: Efficacy and Safety of Oral Sumatriptan Plus Oral Promethazine in Migraine Treatment: a Randomized, Double Blind Clinical Trial
Brief Title: Efficacy and Safety of Oral Sumatriptan Plus Oral Promethazine in Migraine Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shadi Asadollahi, Research Assistant of Neurology, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SB-045
Record Dates: First submitted 2013-03-14; First posted 2013-03-19 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2013-07

CONDITIONS: Migraine With Aura; Migraine Without Aura
MeSH Terms: conditions — Migraine with Aura; Migraine without Aura

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sumatriptan+promethazine (SPr) (Active Comparator): The SPr group denote patients receiving oral sumatriptan (50 mg) plus oral promethazine (50 mg).
  Interventions: Drug: Sumatriptan+Promethazine (SPr)
- Sumatriptan+placebo (SP) (Placebo Comparator): The SP group denote patients receiving oral sumatriptan (50 mg) plus tablet of placebo matched to promethazine.
  Interventions: Drug: Sumatriptan+Promethazine (SPr)

INTERVENTIONS:
Drug: Sumatriptan+Promethazine (SPr)

SUMMARY:
The purpose of this study is to show the efficacy of promethazine in management of patients with moderate to severe migraine

ELIGIBILITY:
Inclusion Criteria:

* Patients who aged 18 to 65 years with a clinical history of migraine with or without aura (International Headache Society categories 1.1 or 1.2) for at least 1 year
* Subjects who have mean frequency of 2-8 migraine attacks per month.

Exclusion Criteria:

* Complex form of migraine, medication overuse headache, history of chronic tension-type headache, ophthalmoplegic, basilar and hemiplegic migraine
* Uncontrolled hypertension (diastolic blood pressure >95 mm Hg or systolic blood pressure >160 mm Hg)
* History or clinical evidence of cerebrovascular or cardiovascular disorder
* Renal impairment or dialysis dependence
* Serious illness (physical or psychiatric disorders)
* Drugs and alcohol abuse
* Pregnancy and breastfeeding
* Allergy or hypersensitivity to promethazine or triptans
* Concurrent use of ergotamine-containing drugs, monoamine oxidize inhibitors, antidepressant, lithium

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Complete headache relief | At 2 hours after first dose
  The primary endpoint variable was the proportions of patients reporting complete headache relief 2 hours after dosing.

SECONDARY OUTCOMES:
Complete headache relief | At 0.5 hour, 1 hour, and 4 hours after first dose
  The secondary endpoint variable was the proportions of patients reporting complete headache relief 0.5 hour, 1 hour, and 4 hours after dosing.
Headache improvement. | At 0.5 hour, 1 hour, 2 hours, 4 hours after first dose.
  The secondary endpoint variable was the proportion of patients experiencing headache improvement at 0.5 hour, 1 hour, 2 hours, 4 hours after dosing.
Using the second dose of study medications. | At 2-48 hours after first dose.
  The secondary endpoint variable was the use of second dose when the severity of headache was still moderate or severe after the first dose within 2-48 hours
Using rescue medication between 2 and 48 hours postdose | At 4-48 hours after second dose.
  The secondary endpoint variable was the use of rescue medication (excluding triptans, and ergot-containing medication) within 4-48 hours after the second dose when headache severity was still at grade 2 ⁄ 3.
Rate of headache recurrence | At 2-48 hours after first dose.
  The secondary endpoint variable was a return to moderate or severe pain within 48 hours of first dose subsequent to primary improvement to mild or no pain at 2 hours.
Occurrence of adverse events. | At 4 hours after first dose.
  Presence or absence of adverse events occurred 4 hours after first dosing.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Emam Hossein Hospital, Tehran, Tehran Province, Iran